CLINICAL TRIAL: NCT05297604
Title: Non-Invasive Intravascular Laser Irradiation Of Blood In The Treatment Of Children With Temporomandibular Disorders - Study Protocol For A Randomized, Controlled, Blind, Clinical Trial
Brief Title: Non-Invasive Intravascular Laser Irradiation Of Blood In The Treatment Of Children With Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMDChildren
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the placeb group will be treated in the same way as the active laser group. The person in charge of the application will simulate the irradiation with the equipment kept off, so that the participant does not identify the group to which he/she belongs to, and the device activation sound (beep) will be turned on at the time of application.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VPBM group (vascular photobiomodulation) (Active Comparator): The participants received a single session of VPBM.
  Interventions: Radiation: Vascular photobiomodulation (VPBM)
- Sham group (simulated vascular photobiomodulation) (Placebo Comparator): The participants received the same treatment as the VPBM group, but the equipment was switched off. To ensure blinding, the sound of the device (beep) was activated at the time of simulated PBM using a telephone.
  Interventions: Radiation: Sham group (simulated vascular photobiomodulation)

INTERVENTIONS:
Radiation: Vascular photobiomodulation (VPBM) — The participants received a 20-minute single session of VPBM. This noninvasive method involves the use of low-power laser coupled to a bracelet designed to transport the light beam transcutaneously over the radial artery. The laser device (DMC Therapy Ec) delivered irradiation with a power of 100 ± 20 mW, wavelength of 660 ± 10 nm (red light) and energy of 120 J applied continuously, with irradiance of 35 W/cm².
  Arms: VPBM group (vascular photobiomodulation)
Radiation: Sham group (simulated vascular photobiomodulation) — Simulated radiation. The participants received a single session.
  Arms: Sham group (simulated vascular photobiomodulation)

SUMMARY:
This study is blind, randomized controlled and have been carried out on children between 6 and 9 years of age, at the Catholic University of Uruguay, Faculty of Health Sciences, Postgraduate School, and surrounding schools. Patients who present temporomandibular disorders, based on the diagnostic criteria will be the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) were included. The laser used was infrared, power 100 mW ±20%, wavelength 660nm ±10 nm, energy parameter 60J, continuous application. The technique is not invasive, the irradiation point is by continuous and direct transcutaneous application to the radial artery by means of a bracelet that inserts the laser beam. One session has been performed. There was a laser group, a placebo group. Participants in all groups were re-evaluated after the procedure, following the same evaluation procedures used initially, evaluating the effects of ILIB on pain and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (ASA I) age six to nine years with diagnosis of TMD in the mixed dentition phase and with jaw deviation and/or deflection. Deviation is defined as the jaw following a deviated path to one side during opening. Deflection is defined as the jaw following a deviated path without returning to the midline when the mouth is fully opened.

Exclusion Criteria:

* Craniofacial anomalies or genetic syndromes due to the greater probability of the development of TMD associated with the malformation, which could be a confounding variable, malocclusion, use of a dental prosthesis, currently undergoing orthodontic treatment, need for orthognathic surgery or physical therapy due to the potential impact on the results of both the diagnosis and treatment, currently undergoing oncological treatment due to the need to avoid conditions that may exert an influence on the response to the proposed treatment and photosensitivity due to the incompatibility with part of the proposed treatment. Individuals on medications could be included and the medications needed to be recorded in the results.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Change in mouth opening range of motion (following clinical protocol of DC/TMD) | Baseline and immediately after the procedure.
  Vertical movement of the jaw was measured using calibrated digital calipers.

SECONDARY OUTCOMES:
Changes in Pain Evaluation | Baseline and immediately after the procedure.
  Pain was assessed using the VAS, which is an instrument for the subjective assessment of pain. The subject makes a mark along a horizontal line with 0 (absence of pain) printed at one end and 10 (extreme pain) printed at the other end. The patient's mark on the line is recorded in the clinical history for reproduction among observers.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sertaje MRF, Goncalves MLL, Gomes AO, Bruno LH, Fossati AL, Viarengo NO, Santos EM, Sobral APT, Mesquita-Ferrari RA, Fernandes KPS, Horliana ACRT, Motta LJ, Bussadori SK. Vascular photobiomodulation in the treatment of children with temporomandibular disorders: Study protocol for a randomized, controlled, blind, clinical trial. Medicine (Baltimore). 2022 Oct 21;101(42):e31228. doi: 10.1097/MD.0000000000031228. PMID 36281107